CLINICAL TRIAL: NCT06891599
Title: Advanced Coagulation Diagnostics Using ROTEM and Standard Coagulation Tests in Hospitalized Patients With Sepsis or Trauma - A Prospective Observational Study (ROSTIC - ROTEM for Sepsis and Trauma Induced Coagulopathy)
Brief Title: ROTEM in Sepsis Trauma Outcome in Intensive Care
Acronym: ROSTIC
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-07157-01; FoUI-985360 (Other Grant/Funding Number: Region Stockholm ALF)
Record Dates: First submitted 2025-03-12; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Sepsis - to Reduce Mortality in the Intensive Care Unit; Trauma Coagulopathy
Keywords: Sepsis; ROTEM; Trauma; Coagulopathy
MeSH Terms: conditions — Sepsis; Wounds and Injuries; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Trauma: Trauma alarm activated at hospital admission New Injury Severity Score (NISS) > 15 Transfer to hospital within 7 days of trauma with NISS > 15
- Sepsis: Meeting Sepsis-3 criteria Receipt of intravenous beta-lactam or aminoglycoside antibiotics within 48 hours of admission
- Control: Patients undergoing elective surgery without expected coagulopathy

SUMMARY:
This prospective observational study aims to investigate the ability of advanced ROTEM analysis using Principal Component Analysis (PCA) to detect early signs of disseminated intravascular coagulation (DIC) and trauma-induced coagulopathy (TIC) in hospitalized patients with sepsis or trauma. Standard coagulation tests and ROTEM measurements will be collected and analyzed in relation to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Trauma patients:

Trauma alarm activated at hospital admission New Injury Severity Score (NISS) > 15 Transfer to hospital within 7 days of trauma with NISS > 15

Sepsis patients:

Meeting Sepsis-3 criteria Receipt of intravenous beta-lactam or aminoglycoside antibiotics within 48 hours of admission

Control group:

Patients undergoing elective surgery without expected coagulopathy

Exclusion Criteria:

Trauma patients:

Isolated chronic subdural hematoma No underlying traumatic event despite trauma alarm Age <18 years

Sepsis patients:

Age <18 years

Control patients:

Ongoing anticoagulant treatment Life-threatening illness (ASA IV-V) Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in Stockhiolm Region
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of abnormal coagulation clusters via PCA of ROTEM in trauma and sepsis patients | Through study completion, an average of 2 years
  Detection of abnormal coagulation clusters via PCA of ROTEM in trauma and sepsis patients

CONTACTS AND LOCATIONS:
Locations (1):
- Region Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
At this time, individual participant data (IPD) will not be shared due to privacy concerns, ethical considerations, and regulatory restrictions. The study involves sensitive patient data, including coagulation profiles and clinical outcomes, which are subject to strict data protection laws and institutional guidelines within Region Stockholm.
  Additionally, data will be pseudoanonymized and stored on secure research servers, with access limited to the study team. While aggregate results will be published in peer-reviewed journals, sharing of raw IPD requires specific ethical and legal approvals, which are not currently in place for unrestricted access.
  However, data access requests for collaborative research may be considered on a case-by-case basis, subject to approval by the relevant ethics committees and data protection authorities.